CLINICAL TRIAL: NCT00948285
Title: Breast Cancer Staging MAgnetic Resonance for Treatment (B-SMART)
Brief Title: Importance of Magnetic Resonance Imaging (MRI) in Treating Breast Cancer
Acronym: BSMART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult accrual
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A09-3519
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; magnetic resonance imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI (Experimental): Preoperative staging with mammogram, ultrasound, and MRI, followed by surgery (n=200)
  Interventions: Procedure: MRI
- Non-MRI (No Intervention): Preoperative staging with mammogram and ultrasound alone, followed by surgery (n=200)

INTERVENTIONS:
Procedure: MRI — magnetic resonance imaging (MRI)
  Arms: MRI

SUMMARY:
The purpose of this study is to determine if the use of magnetic resonance imaging (MRI) for breast cancer translates into better surgical outcomes. MRIs may help ensure that as little healthy tissue is removed as is possible and may help prevent the need for additional surgical procedures.

DETAILED DESCRIPTION:
We propose that the role of preoperative staging-MRI in breast cancer be studied by following the occurrence of negative margins at first surgery and the volume of resection in a randomized prospective study. The need for re-excision is an objective marker of satisfactory local surgery and is available as soon as the final pathology report is back. We propose that the closest margin and the rate of re-excision be used as the primary outcome measures to evaluate the contribution of MRI. In addition, since cosmetic preservation is one of the goals of breast conservation, we propose that cosmetic outcome be used as the secondary outcome measure. The visual analogue scale for cosmetic outcome varies between observers and with time; however, the volume of tissue that is excised is an objective surrogate of cosmetic outcome.15 Since the excised volume is dictated by the tumor volume, the only variable under the surgeon's control is the volume of benign tissue excised in order to obtain negative margins. Hence, in this study, we propose to use a volume index of excised margins as an outcome measure for cosmesis. The index value will be calculated for each subject by adding the two measurements of benign margin for each of the three dimensions measured and multiplying them to produce a volume index for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer patients
* Breast cancer patients identified as conservation candidates by their surgeons

Exclusion Criteria:

* Patients with a history of prior breast cancer treatment (recurrence)
* Patients with breast cancer diagnosis during pregnancy (women who could bear children must have a negative pregnancy test before beginning this study)
* Patients with documented sensitivity to gadolinium (contrast agent used during MRI)
* Patients who weigh more than 350 pounds (weight limit on MRI machine)
* Patients who receive neoadjuvant chemotherapy
* Patients with renal insufficiency (serum Cr > 1.5) due to the danger of nephrogenic systemic sclerosis with the administration of Gadolinium

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-07; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
A difference of 10% in the margin revision rate in women undergoing breast conservation for cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rakhshanda L Rahman, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas, United States